CLINICAL TRIAL: NCT06290544
Title: Cardiovascular Risk Assessment in a Cohort of Italian Patients With Type 1 Diabetes Mellitus - CARDT1
Brief Title: Cardiovascular Risk Assessment in a Cohort of Italian Patients With Type 1 Diabetes Mellitus (CARDT1)
Acronym: CARDT1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCM 1552
Record Dates: First submitted 2023-03-30; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 1; Cardiovascular Diseases
Keywords: Diabetes; Diabetes Mellitus, Type 1; Cardiovascular risk; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cardiovascular Diseases; Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective collection of data with diagnostic procedures different from standard clinical care in a specific cohort of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Other): Subjects with type 1 diabetes mellitus who meet all the inclusion and none exclusion criteria
  Interventions: Other: Standard of care plus additional examinations

INTERVENTIONS:
Other: Standard of care plus additional examinations — The patient will undergo good clinical practice examinations according to guidelines plus The patient will undergo to the evaluation of endothelial dysfunction with ENDOPAT 2000 and whole blood sampling for future omics studies

SUMMARY:
This is a multicenter prospective collection of data with diagnostic procedures different from standard clinical care in a specific cohort of patients, aimed to evaluate cardiovascular risk stratification with the European Society of Cardiology (ESC)/European Association for the Study of Diabetes (EASD) guidelines and "The Steno Type 1 Risk Engine" algorithm. The correlation between CVD risk, atherosclerosis, and microvascular complications of diabetes (retinopathy, nephropathy, and neuropathy) will then be evaluated, and the impact of glycemic variability and other glucose metrics on vascular damage will be characterized. The investigators plan to enroll at least 200 consecutive type 1 diabetes mellitus (T1DM) patients who meet all the inclusion criteria and none of exclusion criteria.

DETAILED DESCRIPTION:
Patients with type 1 diabetes mellitus will be identified in the electronic medical records, and their clinical, anthropometric, and laboratory data, including markers of glycemic variability and other blood glucose metrics, will be collected. Cardiovascular risk will then be assessed using the stratification proposed by ESC/EASD and The Steno Type 1 Risk Engine.

As suggested by the guidelines, according to cardiovascular risk, participants will perform a coronary CT scan in order to investigate coronary anatomy, to study the atherosclerotic plaque morphology, to assess high-risk plaque characteristics, and in case of obstructive coronary artery disease, to investigate myocardial perfusion by adenosine infusion to assess both ischemia and microcirculation dysfunction. Noninvasive B-mode ultrasonography of the supra-aortic trunks will assess for signs of carotid atherosclerosis (i.e., carotid intima media thickness - c-IMT - and carotid plaques). Ankle-arm index (ABI), a noninvasive cardiovascular bio-marker, will provide information on peripheral arterial disease. Endothelial function will be also assessed using the ENDO-PAT 2000 instrument which measures endothelial dysfunction with a peripheral arterial tone detection method.

For the purpose of assessing participants' nutritional habits, participants will be asked to complete the Food Frequency Questionnaire (FFQ) the week prior the visit; once the FFQ will be completed an interview with the nutritionist will be scheduled in order to review and to ascertain its completeness; in addition, the PREDIMED questionnaire for calculating the Mediterranean Diet Adherence Screener score (MEDAS) will be administered to assess adherence to the Mediterranean diet.

An interview with the psychologist will be planned. During that visit the participant will receive information about the rationale of the study regarding psychological aspects, the questionnaires that will be administered and how to fill them out correctly online via the Qualtrics EU platform. The Iowa Gambling Task (IGT) test will then be administered.

Finally, biological samples will be collected for future genomic and epigenetic analyses associated with different cardiovascular disease (CVD) phenotypes and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus.
* Age ≥ 18 years.
* Signed Informed consent

Exclusion Criteria:

* Age < 18 years.
* Pregnancy in progress.
* Type 2 diabetes mellitus.
* Secondary diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Stratify cohort of type 1 diabetes patient according to ESC/EASD 2019 guidelines. | 5 years
  Evaluation of cardiovascular risk class for type 1 diabetic patients using ESC/EASD stratification according to disease duration
Stratify cohort of type 1 diabetes patient according to the Steno Type 1 Risk Engine (ST1RE). | 5 years
  Evaluation of cardiovascular risk class for type 1 diabetic patients using The Steno Type 1 Risk Engine algorithm
Prevalence of cardiovascular disease in type 1 diabetes patients | 5 years
  Prevalence of cardiovascular disease in T1DM cohort defined as one of the following:
  * acute mycardial infarction
  * ischemic stroke
  * peripheral artery disease
  * coronary, carotid or peripheral artery revascularization
  * presence of clinically significant stenosis in coronary CT and/or in carotid ultrasound assessment.

SECONDARY OUTCOMES:
Prevalence of diabetic retinopathy | 5 years
  Prevalence of diabetic retinopathy
Prevalence of diabetic nephropathy | 5 years
  Prevalence of diabetic nephropathy
Prevalence of diabetic neuropathy | 5 years
  Prevalence of diabetic neuropathy
CT-derived calcium score | 5 years
  CT-derived calcium score
Carotid intima-media thickness | 5 years
  Carotid intima-media thickness
Prevalence of endothelial dysfuntion (evaluated using peripheral arterial tone detection method) | 5 years
  Prevalence of endothelial dysfuntion (evaluated using peripheral arterial tone detection method)
Stratify type 1 patient cohort by Food Frequency Questionnaire (FFQ) | At enrollment
  Stratify type 1 patient cohort by Food Frequency Questionnaire (FFQ)
Stratify type 1 patient cohort by the Mediterranean Diet Adherence Screener score (MEDAS) | At enrollment
  Stratify type 1 patient cohort by the Mediterranean Diet Adherence Screener score (MEDAS)
Stratify type 1 patient cohort by psychological profiles using psychological validated questionnaires. | 5 years
  Stratify type 1 patient cohort by psychological profiles using psychological validated questionnaires.
Stratify type 1 patient cohort by lipid profile | 5 years
  Stratify type 1 patient cohort by lipid profile
Stratify type 1 patient by glucose control using HbA1c and Ambulatory Glucose Profile metrics. | 5 years
  Stratify type 1 patient by glucose control using HbA1c and Ambulatory Glucose Profile metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Genovese, MD, Principal Investigator — IRCCS Centro Cardiologico Monzino
Locations (2):
- Italy (2):
  - IRCCS Centro Cardiologico Monzino, Milan
  - Policlinico di Monza, Monza